CLINICAL TRIAL: NCT03204630
Title: Functional Evaluation of Two Infant Formula Supplemented With Probiotics Isolated From Breast Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Collaborators: Maimónides Biomedical Research Institute of Córdoba (Other); Andaluz Health Service (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: P024
Record Dates: First submitted 2016-08-11; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2016-08

CONDITIONS: Infant Nutrition
Keywords: infant nutrition; probiotic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bifido (Active Comparator): Infant formula containing Bifidobacterium breve CECT7263
  Interventions: Dietary Supplement: Bifido
- Lfer (Active Comparator): Infant formula containing Lactobacillus fermentum CECT5716
  Interventions: Dietary Supplement: Lfer
- Control (Placebo Comparator): Standard infant formula
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Lfer — Probiotic bacteria originally isolated from breast milk: the strain Lactobacillus fermentum CECT5716
  Arms: Lfer
Dietary Supplement: Bifido — Probiotic bacteria originally isolated from breast milk: the strain Bifidobacterium breve CECT7263
  Arms: Bifido
Other: Control — Standard infant formula
  Arms: Control

SUMMARY:
A randomized double blinded controlled study including infants at the age of 1 month . Infants are assigned randomly to either infant formula supplemented with B. breve CECT7263 or L.fermentum CECT5716 (Probiotic groups), or the same formula without the probiotic strain (Control group). The primary outcome of the study is the body weight gain of infants. Secondary outcomes are incidence of infections, symptoms related with intestinal function, and fecal microbiota

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants at term (37-42 weeks gestational age) healthy during the first month of life, for reasons unrelated to the study, abandon breastfeeding during the first month of life.
* Signature of informed parental or guardian consent.

Exclusion Criteria:

* Allergic to the protein in cow's milk.
* Lactose intolerant.
* Suffering from a serious metabolic disease.
* They have experienced or are experiencing some severe gastrointestinal disease.
* Receive some form of chronic medication or are receiving antibiotics at the time of capture.
* Low expectation of compliance with the study protocol.
* allergic to any group of antibiotics.

Ages: 3 Weeks to 5 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 236 (Actual)
Dates: Start 2011-01; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Body weight gain | 12 months versus baseline
  Body weight gain at 12 months (grams)

SECONDARY OUTCOMES:
Length | 1,2,4,6,9 and 12 months of age
  Length (cm)
Body weight | 1,2,4,6,9 and 12 months of age
  Body weight of infants at different times (kg)
Incidence of infections | total incidence during intervention (11 months)
  Events of infections diseases during intervention period (Incidence rate)
Bacterial load in feces | 1,2,4,6,9 and 12 months of age
  Counts of Lactobacillus, bifidobacteria, bacteroides, clostridium (CFU/g feces)
Regurgitation | each 2 weeks until 6 months of age and monthly until 12 months of age
  Measurement by score: 1 = not at all, 2 = regurgitation of small amounts during or shortly after feeding, 3 = larger regurgitation during or shortly after feeding, 4 = minor vomiting with time-lag to prior feeding, and 5 = severe vomiting with considerable loss of fluid.
Fecal deposition | each 2 weeks until 6 months of age and monthly until 12 months of age
  Measurement by score:1 = <1 time, 2 = 1-3, 3 = 4-6, 4 = 7-10, and 5 = >10.
Infant colic | each 2 weeks until 6 months of age and monthly until 12 months of age
  Average crying hours per day during the last two days of each period of measurement which is each 2 weeks until 6 months of age and monthly until 12 months of age. Score: no crying; < 3 hours/day;⁯ 3-6 hours/day;⁯ 6-12 hours/day;⁯ > 12 hours/day
Flatulency | each 2 weeks until 6 months of age and monthly until 12 months of age
  Average of duration of flatulence episodes (hours per day) during the last two days of each period of measurement which is each 2 weeks until 6 months of age and monthly until 12 months of age.Measurement by the score:no flatulency; < 3 hours/day;⁯ 3-6 hours/day;⁯ 6-12 hours/day;⁯ > 12 hours/day
Hours of night sleep | each 2 weeks until 6 months of age and monthly until 12 months of age
  Average of time of night sleep (hours per day) during the last two days of each period of measurement which is each 2 weeks until 6 months of age and monthly until 12 months of age.Measurement by the score:⁯ < 4 hours ; 4-6 hours;⁯ 6-9 hours;⁯ 9-12 hours;⁯ > 12 hours
Total hours of sleep/day | each 2 weeks until 6 months of age and monthly until 12 months of age
  ⁯Average of total time of sleep (hours per day) during the last two days of each period of measurement which is each 2 weeks until 6 months of age and monthly until 12 months of age.Measurement by the score:⁯ < 11 hours; ⁯ 11-14 hours; 14-17 hours; 17-20 hours; ⁯ > 20 hours

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Reina Sofía, Córdoba
  - Servicio Andaluz de Salud, Granada

REFERENCES:
- [Derived] Maldonado J, Gil-Campos M, Maldonado-Lobon JA, Benavides MR, Flores-Rojas K, Jaldo R, Jimenez Del Barco I, Bolivar V, Valero AD, Prados E, Penalver I, Olivares M. Evaluation of the safety, tolerance and efficacy of 1-year consumption of infant formula supplemented with Lactobacillus fermentum CECT5716 Lc40 or Bifidobacterium breve CECT7263: a randomized controlled trial. BMC Pediatr. 2019 Oct 21;19(1):361. doi: 10.1186/s12887-019-1753-7. PMID 31630683